CLINICAL TRIAL: NCT05654506
Title: A Multi-center Open-label Trial Evaluating the Efficacy and Safety of Daratumumab SC in Treatment of Patients With Proliferative Glomerulonephritis With Monoclonal Immunoglobulin Deposits (PGNMID)
Brief Title: Daratumumab for Treatment of Proliferative Glomerulonephritis With Monoclonal Immune Deposits
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Fernando Fervenza, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-002587
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-06

CONDITIONS: Proliferative Glomerulonephritis With Monoclonal IgG Deposits
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daratumumab treatment in PGNMID (Experimental): Subjects with native kidney biopsy consistent with membranoproliferative glomerulonephritis with monoclonal immunoglobulin deposits will receive daratumumab.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — 1800 mg subcutaneous (SC) injection (total amount 15 mL) into the right/left abdominal area once weekly for 8 doses followed by once every 2 weeks for an additional 8 doses

SUMMARY:
The purpose of this research is to study the safety and efficacy of daratumumab in inducing complete or partial remission in people with proliferative glomerulonephritis with monoclonal immunoglobulin deposits (PGNMID).

ELIGIBILITY:
Inclusion Criteria:

* Renal biopsy read at Mayo Clinic confirming the diagnosis of PGNMID
* Proteinuria ≥ 1000 mg over 24 hours
* Creatinine clearance ≥ 20 mL/min/SA
* Subjects able and willing to give informed consent
* For female subjects of reproductive childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously during the Treatment Period, during any dose interruptions, and for 3 months after the last dose of any component of the treatment regimen. Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. This birth control method must include one highly effective form of contraception (tubal ligation, intrauterine device, hormonal [birth control pills, injections, hormonal patches, vaginal rings, or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin 4 weeks prior to dosing. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy or bilateral oophorectomy

  * A woman of childbearing potential must have 2 negative serum or urine pregnancy tests at Screening, first within 10 to 14 days prior to dosing and the second within 24 hours prior to dosing.
  * A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 3 months after receiving the last dose of any component of the treatment regimen.
* For male subjects of reproductive potential who are sexually active with females of

  * reproductive potential must always use a latex or synthetic condom during the study and for 3 months after discontinuing study treatment (even after a successful vasectomy).
  * Male subjects of reproductive potential must not donate sperm during the study or for 3 months after the last dose of study treatment.
  * Must sign an informed consent form (ICF) or their legally acceptable representative must sign indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.

Exclusion Criteria:

* Pregnant or planning to become pregnant
* Seropositive for human immunodeficiency virus (HIV)
* Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) will also be excluded. Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR and can be included.
* Multiple myeloma defined as >10% plasma cells on bone marrow biopsy and M-spike > 3 g/dL and presence of myeloma defining event (hypercalcemia, cast nephropathy, bone disease, or anemia), or plasma cells >60% or FLC ratio of involved to uninvolved > 100
* Abnormal clinical labs defined as: anemia with Hgb < 8.0 g/dL, thrombocytopenia with platelet count < 75,000, leukopenia with WBC < 3.5, or neutropenia with ANC < 1000, AST/ALT > 2.5 X ULN, bilirubin > 2 X ULN
* Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is < 50% of predicted normal.
* Moderate or severe persistent asthma withing the past 2 years or uncontrolled asthma of any classification. Note the participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate.
* Clinically significant cardiac disease including:

  * Myocardial infarction within 6 months before randomization, or unstable or uncontrolled disease/condition related to cardiac dysfunction (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV)
  * Uncontrolled arrythmia
* Prior or current exposure to any of the following:

  * To daratumumab or other anti-CD-38 therapies (unless a re-treatment study)
  * Exposure to an investigational drug (including investigational vaccine) or invasive investigational medical device for any indication within 4 weeks or 5 pharmacokinetic half-lives, whichever is longer.
  * Focal radiation therapy within 14 days prior to randomization with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complication
* Unable to provide consent
* Patients receiving therapy with oral prednisone or glucocorticoid equivalent in the last 4 weeks. Patients treated with low dose oral prednisone or glucocorticoid are allowed to be included if they are taking the medication for conditions unrelated to PGNMID (e.g., asthma, gout) at a daily dose of 10mg or less.
* Patients who had received immunosuppressive therapy with MMF, cyclosporine, tacrolimus, or azathioprine in the last 3 months. For patients who have shown no reduction in proteinuria despite ≥ 3 months of MMF, AZA, cyclosporine, tacrolimus, etc, are allowed to enter the study after discontinuing these meds for 7 or more days.
* Patients who have received cyclophosphamide or bortezomib will be allowed to participate as long as there is clear evidence of lack of response to cyclophosphamide or bortezomib defined as lack of achieving complete or partial remission.
* Patients who received rituximab previously with CD20 count of < 20 cells/microliter at the time of enrollment
* Have received vaccination with live attenuated vaccines within 4 weeks of first study agent administration
* A history of malignancy (other than multiple myeloma) unless all treatment of that malignancy was completed at least 2 years before consent and the patient has no evidence of disease before the date of randomization. Exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in proteinuria | Baseline, 12 months
  Change in protein in the urine from baseline to 12 months of follow-up

SECONDARY OUTCOMES:
Number of Treatment-Emergent Adverse Events | 12 months
  Number of treatment-emergent adverse events as defined as major infection (defined as those requiring ED visit or hospitalization for development of pneumonia, sepsis, severe UTI or pyelonephritis, meningitis and c.diff infections), grade 3 or 4 anemia, leukopenia, thrombocytopenia, neutropenia or hospitalization due to eye complication.
Proteinuria at 6 Months | 6 months
  Measured using 24 hour urine collection reported in mg/24 h
Serum Albumin at 6 months | 6 months
  Blood serum collected and reported in g/dL
Serum Albumin at 12 months | 12 months
  Blood serum collected and reported in g/dL
Serum Creatinine at 6 Months | 6 months
  Blood serum collected and reported in mg/dL
Serum Creatinine at 12 Months | 12 months
  Blood serum collected and reported in mg/dL
Hematuria at 6 months | 6 months
  Measured by urinalysis (urine testing) reported in red blood cells per high power field (RBC/HPF)
Hematuria at 12 months | 12 months
  Measured by urinalysis (urine testing) reported in red blood cells per high power field (RBC/HPF)
Complete remission status | 12 months
  Number of subjects to achieve complete remission at 12 months defined as < 500 mg proteinuria/24 hours and no than a 15% reduction in GFR as determined by creatinine clearance
Partial remission status | 12 months
  Number of subjects to achieve partial remission status at 12 months defined as > 50% reduction in 24-hour proteinuria and no greater than a 30% reduction in baseline GFR as determined by creatinine clearance
Maintenance of remission | 24 months
  Number of subjects to maintain their remission status at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fervenza, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - University North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials